CLINICAL TRIAL: NCT05973331
Title: Prospective Validation of an EHR-based Model to Predict Pancreatic Cancer Risk Using Multicenter US Data
Brief Title: Prospective Validation of an EHR-based Pancreatic Cancer Risk Model
Status: Active, not recruiting | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Massachusetts Institute of Technology (Other)
Responsible Party: Principal Investigator, Limor Appelbaum, Staff Scientist, Beth Israel Deaconess Medical Center
Other Study IDs: 2023Trial
Record Dates: First submitted 2023-07-17; First posted 2023-08-02 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Pancreatic Adenocarcinoma; Predictive Cancer Model

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- prospective general opulation cohort: Males and females age >= 40 years, without a personal history of PDAC or current PDAC, with at least 2 clinical encounters to the HCO within the year prior to the study start date.
  Interventions: Other: Pancreatic Cancer Risk Model (PRISM)

INTERVENTIONS:
Other: Pancreatic Cancer Risk Model (PRISM) — A neural network model (PrismNN) and a logistic regression model (PrismLR) that use routinely collected EHR data to stratify individuals from the general population into PDAC risk groups

SUMMARY:
The goal of this prospective observational cohort study is to validate a previously developed pancreatic cancer risk prediction algorith (the PRISM model) using electronic health records from the general population. The main questions it aims to answer are:

* Will a pancreatic cancer risk model, developed on routine EHR data, reliably and accurately predict pancreatic cancer in real-time?
* What is the average time from model deployment and risk prediction, to the date of pancreatic cancer development and what is the stage of pancreatic cancer at diagnosis? The risk model will be deployed on data from individuals eligible for the study. Each individual will be assigned a risk score and tracked over time to assess the model's discriminatory performance and calibration.

DETAILED DESCRIPTION:
To prospectively validate, implement in real-time, and assess performance of an EHR- based PDAC risk-prediction model. To test the hypothesis that our model will reliably predict PDAC in a real-time clinical setting, we will conduct a multi-center prospective cohort study, deploying the PDAC risk model within the TriNetX federated network database, and will take the following steps:

i) generate a risk prediction score for each individual under the care of 44 health care organizations (HCOs) in the USA ii) follow all individuals for up to 3 years to assess the primary end-point of PDAC development.

The following metrics will be used to test the discriminative performance and calibration of the EHR-based PDAC risk model in predicting incident PDAC, at the end of the 3-year period:

1. AUROC, sensitivity, specificity, PPV/NPV for assessing discrimination
2. Calibration: for assessing the accuracy of estimates, based on the estimated to observed number of events

ELIGIBILITY:
Inclusion Criteria:

* Male and females age >= 40 years from 44 US HCOs from the TriNetX platform
* at least 2 clinical encounters to the HCO, within the last year, before the study start date

Exclusion Criteria:

* Personal history of PDAC or current PDAC
* Age below 40

Notes on sampling method: no sampling was performed. All eligible individuals are included in this study.

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The cohort will be selected from 44 eligible HCOs comprised of community hospitals, outpatient clinics and academic medical centers from across the US.
Sampling Method: Non-Probability Sample
Enrollment: 6134060 (Actual)
Dates: Start 2023-04-21 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Area under the receiver operating characteristic curve (AUROC) of PRISM for all groups stratified | 6 months from index date
  To assess the discriminatory performance of PRISM for prospective identification of high-risk individuals for PDAC development. ROCs and AUROC numbers will be calculated for the whole population and groups stratified by age, sex, race, and geographical location.
Area under the receiver operating characteristic curve (AUROC) of PRISM for all groups stratified | at 1 year
  To assess the discriminatory performance of PRISM for prospective identification of high-risk individuals for PDAC development. ROCs and AUROC numbers will be calculated for the whole population and groups stratified by age, sex, race, and geographical location.
Area under the receiver operating characteristic curve (AUROC) of PRISM for all groups stratified | at 2 years
  To assess the discriminatory performance of PRISM for prospective identification of high-risk individuals for PDAC development. ROCs and AUROC numbers will be calculated for the whole population and groups stratified by age, sex, race, and geographical location.
Area under the receiver operating characteristic curve (AUROC) of PRISM for all groups stratified | at 3 years
  To assess the discriminatory performance of PRISM for prospective identification of high-risk individuals for PDAC development. ROCs and AUROC numbers will be calculated for the whole population and groups stratified by age, sex, race, and geographical location.
Calibration of PRISM for all groups stratified | 6 months from index date
  To access how well the risk prediction by PRISM aligns with observed risk without recalibration. Calibration plots will be created for the whole population and groups stratified by age, sex, race, and geographical location.
Calibration of PRISM for all groups stratified | at 1 year
  To access how well the risk prediction by PRISM aligns with observed risk without recalibration. Calibration plots will be created for the whole population and groups stratified by age, sex, race, and geographical location.
Calibration of PRISM for all groups stratified | at 2 years
  To access how well the risk prediction by PRISM aligns with observed risk without recalibration. Calibration plots will be created for the whole population and groups stratified by age, sex, race, and geographical location.
Calibration of PRISM for all groups stratified | at 3 years
  To access how well the risk prediction by PRISM aligns with observed risk without recalibration. Calibration plots will be created for the whole population and groups stratified by age, sex, race, and geographical location.
PRISM performance metrics of high-risk group for direct screening | 6 months from index date
  To evaluate sensitivity, specificity, PPV, and SIR for patients identified as high-risk by PRISM. Numbers will be calculated for the whole population and groups stratified by age, sex, race, and geographical location. Risk threshold determined based on Standardized Incidence Ratio of 5 or greater. The absolute one-year risk thresholds are 0.1834% for PrismNN and 0.2048% risk for PrismLR. SIR 5 or greater was chosen because it is comparable to the current screening inclusion threshold for individuals with an inherited predisposition.
PRISM performance metrics of high-risk group for direct screening | at 1 year
  To evaluate sensitivity, specificity, PPV, and SIR for patients identified as high-risk by PRISM. Numbers will be calculated for the whole population and groups stratified by age, sex, race, and geographical location. Risk threshold determined based on Standardized Incidence Ratio of 5 or greater. The absolute one-year risk thresholds are 0.1834% for PrismNN and 0.2048% risk for PrismLR. SIR 5 or greater was chosen because it is comparable to the current screening inclusion threshold for individuals with an inherited predisposition.
PRISM performance metrics of high-risk group for direct screening | at 2 years
  To evaluate sensitivity, specificity, PPV, and SIR for patients identified as high-risk by PRISM. Numbers will be calculated for the whole population and groups stratified by age, sex, race, and geographical location. Risk threshold determined based on Standardized Incidence Ratio of 5 or greater. The absolute one-year risk thresholds are 0.1834% for PrismNN and 0.2048% risk for PrismLR. SIR 5 or greater was chosen because it is comparable to the current screening inclusion threshold for individuals with an inherited predisposition.
PRISM performance metrics of high-risk group for direct screening | at 3 years
  To evaluate sensitivity, specificity, PPV, and SIR for patients identified as high-risk by PRISM. Numbers will be calculated for the whole population and groups stratified by age, sex, race, and geographical location. Risk threshold determined based on Standardized Incidence Ratio of 5 or greater. The absolute one-year risk thresholds are 0.1834% for PrismNN and 0.2048% risk for PrismLR. SIR 5 or greater was chosen because it is comparable to the current screening inclusion threshold for individuals with an inherited predisposition.
PRISM performance metrics of medium-risk group for biomarker testing | 6 months from index date
  To evaluate sensitivity, specificity, PPV, and SIR for patients identified as medium-risk by PRISM. Numbers will be calculated for the whole population and groups stratified by age, sex, race, and geographical location. Risk threshold determined by specificity 85%, with sensitivity around 46%. The absolute one-year risk thresholds are 0.0574% for PrismNN and 0.0564% for PrismLR. Prism operates as a tiered system for identifying individuals in need of screening with this lower risk threshold.
PRISM performance metrics of medium-risk group for biomarker testing | at 1 year
  To evaluate sensitivity, specificity, PPV, and SIR for patients identified as medium-risk by PRISM. Numbers will be calculated for the whole population and groups stratified by age, sex, race, and geographical location. Risk threshold determined by specificity 85%, with sensitivity around 46%. The absolute one-year risk thresholds are 0.0574% for PrismNN and 0.0564% for PrismLR. Prism operates as a tiered system for identifying individuals in need of screening with this lower risk threshold.
PRISM performance metrics of medium-risk group for biomarker testing | at 2 years
  To evaluate sensitivity, specificity, PPV, and SIR for patients identified as medium-risk by PRISM. Numbers will be calculated for the whole population and groups stratified by age, sex, race, and geographical location. Risk threshold determined by specificity 85%, with sensitivity around 46%. The absolute one-year risk thresholds are 0.0574% for PrismNN and 0.0564% for PrismLR. Prism operates as a tiered system for identifying individuals in need of screening with this lower risk threshold.
PRISM performance metrics of medium-risk group for biomarker testing | at 3 years
  To evaluate sensitivity, specificity, PPV, and SIR for patients identified as medium-risk by PRISM. Numbers will be calculated for the whole population and groups stratified by age, sex, race, and geographical location. Risk threshold determined by specificity 85%, with sensitivity around 46%. The absolute one-year risk thresholds are 0.0574% for PrismNN and 0.0564% for PrismLR. Prism operates as a tiered system for identifying individuals in need of screening with this lower risk threshold.

SECONDARY OUTCOMES:
Timing of incident PDAC occurrence | 6 months from index date
  To evaluate how long in advance before PDAC occurrence should be expected for PRISM models to make high-risk predictions. Distribution plots of the date of PDAC incidence for high/medium-risk groups (defined in Outcome 3 and Outcome 4) will be created.
Timing of incident PDAC occurrence | at 1 year
  To evaluate how long in advance before PDAC occurrence should be expected for PRISM models to make high-risk predictions. Distribution plots of the date of PDAC incidence for high/medium-risk groups (defined in Outcome 3 and Outcome 4) will be created.
Timing of incident PDAC occurrence | at 2 years
  To evaluate how long in advance before PDAC occurrence should be expected for PRISM models to make high-risk predictions. Distribution plots of the date of PDAC incidence for high/medium-risk groups (defined in Outcome 3 and Outcome 4) will be created.
Timing of incident PDAC occurrence | at 3 years
  To evaluate how long in advance before PDAC occurrence should be expected for PRISM models to make high-risk predictions. Distribution plots of the date of PDAC incidence for high/medium-risk groups (defined in Outcome 3 and Outcome 4) will be created.
Tumor stage at PDAC diagnosis | 6 months from index date
  stage at diagnosis per tumor registry/pathology report
Tumor stage at PDAC diagnosis | at 1 year
  stage at diagnosis per tumor registry/pathology report
Tumor stage at PDAC diagnosis | at 2 years
  stage at diagnosis per tumor registry/pathology report
Tumor stage at PDAC diagnosis | at 3 years
  stage at diagnosis per tumor registry/pathology report

CONTACTS AND LOCATIONS:
Overall Officials: Limor Appelbaum, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No